CLINICAL TRIAL: NCT06173804
Title: A Senior Center-Based Multilevel Lifestyle Intervention to Improve Physical Function in Older Adults With Type 2 Diabetes (RESILIENT)
Brief Title: Multilevel Lifestyle Intervention to Improve Physical Function in Older Adults With Type 2 Diabetes
Acronym: RESILIENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000013
Record Dates: First submitted 2023-11-29; First posted 2023-12-18 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Evidence based lifestyle intervention; Older Adults; Physical Function; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A pre-post-test study to assess the implementation outcomes and preliminary health responses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention group (Experimental): The study team will assess improvements in physical function assessed by the short physical performance battery and other health-related measures (diabetes knowledge, self-efficacy, social support, physical activity, diet consumption, HbA1c, and quality of life).
  Interventions: Other: Adapted Look Ahead Lifestyle Intervention

INTERVENTIONS:
Other: Adapted Look Ahead Lifestyle Intervention — Participants will be educated about improving healthy lifestyles involving physical activity and healthy eating to improve physical function and improve glycemic control.
  Other Names: Multilevel Lifestyle Intervention

SUMMARY:
The purpose of this study is to explore strategies to effectively implement senior-center-based multilevel lifestyle interventions adapted from evidence-based lifestyle interventions to promote physical function and quality of life in diverse older adults with Type 2 Diabetes (T2D).

DETAILED DESCRIPTION:
Aim 1: Work with community stakeholders including individuals with T2D, family members, and senior center staff to adapt evidence-based lifestyle interventions, and develop implementation strategies.

Aim 2: Conduct a senior-center-based 6-month pre- and post-pilot study and collect recruitment, enrollment, retention rate, fidelity, program satisfaction and experience, and stakeholder acceptance using quantitative and qualitative data.

Aim 3: Assess the preliminary health-related responses to the intervention in older adults with T2D in the 6-month trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥60 years
2. Self-reported T2D diagnosis with verification from a health report
3. Live within the census tract of the selected senior center, or a member of the senior center
4. No significant cognitive impairment as defined by MMSE (score≥20) (46) which may influence diabetes self-management
5. Can speak and understand either English or Spanish
6. Agree to participate in the study procedures

Exclusion Criteria:

1. Severe chronic conditions without physician's permission to participate (e.g., severe heart disease and end-stage renal disease);
2. Unwillingness to sign the consent form; and
3. Enrollment in other diabetes management programs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting study | Baseline, 3, 6, and 12 months
  Feasibility refers to how feasible to conduct the study. In this study, feasibility will be assessed by data such as participant recruitment, enrollment, education session attendance, and retention rate.
Acceptability | Baseline, 3, 6, and 12 months
  Acceptability refers to how well an intervention will be received by the target population and the extent to which an intervention might meet the needs of the target population. Acceptability will be assessed through qualitative interview with participants to explore their experience, and perceptions with the intervention.

SECONDARY OUTCOMES:
Body Weight | Baseline, 3, 6, and 12 months
  Measured in pounds with participant in light clothes and without shoes
Systolic Blood Pressure | Baseline, 3, 6, and 12 months
  Sitting blood pressure will be measured after at least five minutes of rest.
Diastolic Blood Pressure | Baseline, 3, 6, and 12 months
  Sitting blood pressure will be measured after at least five minutes of rest.
Short Physical Performance Battery (SPPB) | Baseline, 3, 6, and 12 months
  The SPPB is a series of physical tests used to assess a person's lower extremity function. SPPB scores range from zero to 12 possible points. A higher score indicated better physical performance.
Grip Strength | Baseline, 3, 6, and 12 months
  Grip strength will be measured in both hands, and the dominant hand will be recorded.
Glycated Hemoglobin (HbA1c) | Baseline, 3, 6, and 12 months
  HbA1c is a blood test that is used to assess and monitor the average level of glucose over the past two to three months.
Lipid profile | Baseline, 3, 6, and 12 months
  It is a blood test that measures the levels of fats and fatty substances in the blood. The following measurements in the profile will be assessed: cholesterol, LDL (low-density lipoprotein) cholesterol, HDL (high-density lipoprotein) cholesterol, and triglycerides.
IPAQ-12 | Baseline, 3, 6, and 12 months
  This scale contains 12 items that are a self-reported measure of physical activity. Scores are typically expressed in minutes per week. Higher scores indicate higher levels of physical activity, whereas lower scores suggest sedentary or low activity levels.
MoCA | Baseline, 3, 6, and 12 months
  MoCA is a 30-point questionnaire that tests various cognitive domains, including memory, attention, language, abstraction, executive functions, visual skills, calculation, and orientation. The score ranges from 0-30, and higher score indicates better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Du, PhD, MPH, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Health System Texas Diabetic Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The deidentified quantitative data from the 15 participants such as demographics and clinical data could be shared upon request from the applicant after the study findings have been published in peer-reviewed journals.
  The biospecimen collected at the senior center will be transported to the School of Nursing Biobehavioral Laboratory by the laboratory staff or the PI in a dry ice container on the same day of data collection.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data may be shared after peer-reviewed journal publication after study completion or as summary results on ClinicalTrials.gov